CLINICAL TRIAL: NCT03340935
Title: Safety, Feasibility and Metabolic Effects of the Fasting Mimicking Diet (FMD) in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Filippo de Braud (Other)
Collaborators: University of Milan (Other)
Responsible Party: Sponsor-Investigator, Filippo de Braud, Dean of Medical Oncology and Hematology Department, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Organization: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 10/17
Record Dates: First submitted 2017-11-05; First posted 2017-11-14 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Malignant Neoplasm; Cancer
Keywords: fasting mimicking diet; malignant neoplasm; metabolism; metabolic effects; adjuvant treatment; metastatic setting
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fasting mimicking diet (Experimental): Fasting mimicking diet (FMD)
  Interventions: Other: Fasting mimicking diet

INTERVENTIONS:
Other: Fasting mimicking diet — Fasting Mimicking Diet (or FMD) consists in a 5-day plant-based, low-calorie (600 Kcal on day 1, followed by 300 KCal/day on days 2 to 5), low-protein, low carbohydrate diet

SUMMARY:
In preclinical studies, cyclic calorie-restricted diets reduce the risk of several cancers and improve the antitumor activity of standard treatments against already established malignancies.In particular, the fasting mimicking diet (FMD), a plant-based, calorie-restricted, low carbohydrate, low-protein diet to be repeated cyclically every 3-4 weeks, enhances the antitumor activity of cytotoxic chemotherapy, while contemporarily protecting healthy tissues and stimulating antitumor immunity. Most of these effects are likely mediated by the reduction of blood glycemia and growth factors, such as insulin and insulin-like growth factor 1 (IGF-1). When administered to healthy volunteers, cyclic FMD has been shown to be safe and capable of reducing risk factors for different chronic diseases. However, the effects of the FMD in cancer patient populations have not been evaluated so far. This study aims to assess the safety, feasibility and metabolic effects of the FMD in cancer patients treated with different standard antitumor therapies. Patients with any malignancy, with the exception of small cell neuroendocrine tumors, will be considered for enrollment in this study. The FMD will be administered up to a maximum of 8 consecutive cycles in combination with standard adjuvant treatments or therapies for advanced disease.

DETAILED DESCRIPTION:
Tumor and normal cells display differential sensitivity to nutrient and growth factor deprivation. Due to high proliferation rates, most tumor cells depend on continuous energy and metabolic replenishment to renew and duplicate their intracellular components, such as lipid membranes, organelles, DNA and proteins; moreover, as a consequence of constitutive activation of oncogenic pathways, they are unable to halt their proliferation during starvation. This exposes them to acute energetic and anabolic crisis when nutrients (e.g. glucose, amino acids) and growth factors (e.g. insulin) in the extracellular environment are scarce. Starvation-induced toxicity is even higher when tumor cells are exposed to cytotoxic compounds, such as DNA damaging agents. Indeed, repair mechanisms that are essential to survive damage induced by cytotoxic chemotherapy require energy (in the form of ATP units) and metabolic precursors (e.g., nucleotides) that are potentially reduced at the tumor site during nutrient deprivation.

Conversely, cells of healthy tissues are more capable of adapting their proliferation and metabolism to the metabolic contexture. In conditions of nutrient and growth factor deprivation, most normal cells enter a quiescent proliferative status, thus reducing energy- and metabolite-requiring processes, such as DNA, lipid and protein synthesis; they also activate catabolic processes, such as autophagy, which provide the minimal amount of metabolites to survive starvation. Proliferative quiescence not only prevents the occurrence of damage to intracellular structures and orgenelles, but also favors their repair by sparing energy units and essential metabolites.

This differential response to starvation by cancer and normal cells could be potentially exploited to selectively target in vivo human cancers, while sparing healthy tissues. Cyclic fasting or a plant-based, calorie-restricted, low-carbohydrate low-protein diet known as fasting mimicking diet (FMD), are two approaches that have emerged in recent years to selectively target the metabolic vulnerabilities of malignant cells. Indeed, they are capable of inducing meaningful modifications in systemic metabolism, such as reduction of blood glucose insulin and insulin-like growth factor (IGF-1) in both mice and healthy volunteers.

Studies performed in preclinical models of several cancers have demonstrated that cyclic fasting/FMD produce synergistic anticancer effects when combined with cytotoxic chemotherapy, while protecting normal tissues and stimulating antitumor immunity. So far, only a few studies have tested the effects of fasting/FMD in healthy volunteers or cancer patients.

In healthy volunteers, three consecutive cycles of FMD have been shown to be safe and associated with meaningful changes in risk factors for chronic diseases. In cancer patients, a few small studies have demonstrated that short-term fasting (1-3 consecutive days every 3-4 weeks) is feasible and safe in combination with standard chemotherapy, including platinum-based chemotherapy. However, the effects of the FMD in cancer patients have not been investigated so far.

This study,aims to test the safety, feasibility and metabolic effects of the fasting-mimicking diet (FMD) in patients with different malignant neoplasms.

Patients highly motivated to follow the FMD in combination with their standard treatments, will be considered for enrollment in this study. All enrolled patients will be prescribed the same 5-day FMD regimen, which consists of a calorie-restricted (about 600 Kcal on day 1, 300 Kcal/day on days 2 to 5), low-carbohydrate, low-protein diet, which will be repeated every 21-28 days. A maximum of 8 consecutive FMD cycles will be prescribed. During each of the 5 days on FMD, patients will have at least one daily contact (by email or phone) with the study staff to communicate body weight, blood pressure, health conditions, adverse events and the amount of food and beverages introduced (also reported in daily food diaries). In the interval between consecutive FMD cycles, patients will not be prescribed any maintenance diet, but will receive generic dietary recommendations based on World Cancer Research Fund (WCRF 2007) or the American Cancer Society (ACS 2012) recommendations for cancer prevention and cancer survivors.

Patients with any malignancy, except for small cell neuroendocrine tumors, and any disease stage are potentially eligible for this study. Patients with a body mass index (BMI) < 20 kg/m2, as well as patients who lost more than 5% of their basal weight in the last 3 months, will be excluded from the study. Patients with severe comorbidities, or diabetes mellitus requiring pharmacologic therapies, will be also excluded. The FMD will be permanently discontinued in the case of FMD-related grade 4 adverse events (AEs) or serious adverse events (SAEs), or in the case that patient BMI goes below 20 kg/m2 during the FMD and is not restored between two consecutive FMD cycles.

Patients enrolled in this study will receive standard-of-care treatment for their tumor, including chemotherapy, radiotherapy, molecular target therapy, immunotherapy or best supportive care. Both patients with metastatic disease and patients undergoing adjuvant therapy after curative surgery will be candidate to enter this protocol.

The primary endpoint of the study is safety of the FMD in combination with standard antitumor treatments. Safety will be assessed by reporting and grading FMD-related AEs according to NCI Common Terminology Criteria for Adverse Events (CTCAEs) v 4.03. SAEs will be also reported.

FMD feasibility, FMD-induced metabolic effects, weight changes, and modifications of other blood and biochemical parameters will be secondary endpoints.

Feasibility will be assessed by evaluating the patient ability to comply with the prescribed dietary scheme. To do so, all patients will fill a daily food diary during each of the 5 days on FMD. At the end of the study, diaries will be analyzed. Based on the presence of major and minor deviations from the prescribed dietary scheme, patients will be defined as "compliant" or "not compliant".

FMD-induced metabolic effects will be quantified by measuring blood and urine metabolites and growth factors before the initiation and at completion of each FMD cycle (i.e. before resuming the normal diet). Absolute and relative metabolite and growth factor modifications will be reported. Standard metabolites (e.g. blood glucose, triglycerides, total and HDL cholesterol, urine ketone bodies) will be measured. In selected patients, plasma and whole blood fatty acids and some amino acids will be measured too.

The effect of the FMD on patient weight will be assessed by measuring absolute and relative weight changes during each FMD cycle and along with subsequent cycles.

Changes occurring in other blood parameters, including blood cell counts, aspartate and alanine transaminases, blood urea nitrogen, creatinine and uric acid, C reactive protein, total proteins and albumin, will be also measured before and at the end of each FMD cycle.

Finally, diet-induced changes in peripheral blood fatty acid and phospholipid profiles, as well as of immune cell populations, will be assessed in selected patients as exploratory analyses.

ELIGIBILITY:
Inclusion criteria:

* Cytologically or Histologically confirmed diagnosis of malignant neoplasm
* Capability of swallowing plant-based foods foreseen by the FMD
* Body mass index (BMI) ≥ 20 kg/m2
* Adequate bone marrow function, including:

  1. Hemoglobin > 9 g/dl
  2. Piatelets > 75,000/µl
  3. Absolute neutrophil count (ANC) > 1,500/µl
* Creatinine < 1.5 mg/dl or calculated creatinine clearance ≥50 mL/min
* Uric acid < 6 mg/dl
* Fasting glucose > 65 mg/dl
* Total bilirubin < 2 mg/dl or < ULN, except for patients with Gilbert syndrome
* Written informed consent according to the local Ethics Committee requirements
* Willing and ability to accomplish blood and urinary examinations according to the protocol
* Ability to maintain a daily contact (by phone or email) with the study staff for the communication of crucial clinical information, including daily body weight, blood pressure, health status and adverse events during each of the 5 days on diet

Exclusion criteria:

* Small cell neuroendocrine carcinoma
* Unintentional weight loss ≥ 5% in the last 3-6 months
* Known HIV infection
* Pregnancy or lactation
* History of alcohol abuse
* Diagnosis of diabetes mellitus type I or type II that requires medical treatment
* Fasting glucose > 200 mg/dl
* Clinically meaningful cardiovascular, renal or pulmonary diseases
* Current treatment with antipsychotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Safety of the fasting mimicking diet (FMD) in cancer patients | 2 years
  Safety is assessed by recording each adverse (AE) occurring during the period on diet. All AEs will be graded according to the NCI CTCAE v 4.03. Serious adverse events (SAEs) will be also reported.

SECONDARY OUTCOMES:
Feasibility of the FMD in cancer patients | 16 months
  Feasibility is defined as the ability of the patient to comply with the prescribed dietary regimen. It will be assessed through the analysis of food diaries filled by patients during the five days of each FMD cycle.
Metabolic effects of the FMD | 16 months
  FMD-induced metabolic changes will be evaluated by measuring blood metabolites (glucose, cholesterol, triglycerides) and urinary ketone bodies before and at the completion of each FMD cycle.
Effects of the FMD on blood growth factors | 16 months
  FMD-induced changes in blood growth factors will be evaluated by measuring modifications of plasma insulin and serun insulin-like growth factor 1 (IGF-1) concentration before and at the completion of each FMD cycle
Weight changes during the FMD | 16 months
  Percent changes in body weight will be measured during each FMD cycle and across subsequent FMD cycles.
Changes in blood cell counts | 16 months
  FMD-induced changes in blood cell counts
Changes in kidney function parameters. | 16 months
  FMD-induced changes in parameters linked to kidney function, such as blood urea nitrogen, creatinine and uric acid.
Changes in liver parameters | 16 months
  FMD-induced changes in parameters linked to liver function, such as aspartate and alanine transaminases, total bilirubin.

CONTACTS AND LOCATIONS:
Overall Officials: Filippo de Braud, M.D., Principal Investigator — SC Oncologia Medica 1, Fondazione IRCCS Istituto Nazionale dei Tumori
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vernieri C, Casola S, Foiani M, Pietrantonio F, de Braud F, Longo V. Targeting Cancer Metabolism: Dietary and Pharmacologic Interventions. Cancer Discov. 2016 Dec;6(12):1315-1333. doi: 10.1158/2159-8290.CD-16-0615. Epub 2016 Nov 21. PMID 27872127
- [Result] Brandhorst S, Choi IY, Wei M, Cheng CW, Sedrakyan S, Navarrete G, Dubeau L, Yap LP, Park R, Vinciguerra M, Di Biase S, Mirzaei H, Mirisola MG, Childress P, Ji L, Groshen S, Penna F, Odetti P, Perin L, Conti PS, Ikeno Y, Kennedy BK, Cohen P, Morgan TE, Dorff TB, Longo VD. A Periodic Diet that Mimics Fasting Promotes Multi-System Regeneration, Enhanced Cognitive Performance, and Healthspan. Cell Metab. 2015 Jul 7;22(1):86-99. doi: 10.1016/j.cmet.2015.05.012. Epub 2015 Jun 18. PMID 26094889
- [Result] de Groot S, Vreeswijk MP, Welters MJ, Gravesteijn G, Boei JJ, Jochems A, Houtsma D, Putter H, van der Hoeven JJ, Nortier JW, Pijl H, Kroep JR. The effects of short-term fasting on tolerance to (neo) adjuvant chemotherapy in HER2-negative breast cancer patients: a randomized pilot study. BMC Cancer. 2015 Oct 5;15:652. doi: 10.1186/s12885-015-1663-5. PMID 26438237
- [Result] Di Biase S, Lee C, Brandhorst S, Manes B, Buono R, Cheng CW, Cacciottolo M, Martin-Montalvo A, de Cabo R, Wei M, Morgan TE, Longo VD. Fasting-Mimicking Diet Reduces HO-1 to Promote T Cell-Mediated Tumor Cytotoxicity. Cancer Cell. 2016 Jul 11;30(1):136-146. doi: 10.1016/j.ccell.2016.06.005. PMID 27411588
- [Result] Dorff TB, Groshen S, Garcia A, Shah M, Tsao-Wei D, Pham H, Cheng CW, Brandhorst S, Cohen P, Wei M, Longo V, Quinn DI. Safety and feasibility of fasting in combination with platinum-based chemotherapy. BMC Cancer. 2016 Jun 10;16:360. doi: 10.1186/s12885-016-2370-6. PMID 27282289
- [Result] Lee C, Raffaghello L, Brandhorst S, Safdie FM, Bianchi G, Martin-Montalvo A, Pistoia V, Wei M, Hwang S, Merlino A, Emionite L, de Cabo R, Longo VD. Fasting cycles retard growth of tumors and sensitize a range of cancer cell types to chemotherapy. Sci Transl Med. 2012 Mar 7;4(124):124ra27. doi: 10.1126/scitranslmed.3003293. Epub 2012 Feb 8. PMID 22323820
- [Result] Safdie FM, Dorff T, Quinn D, Fontana L, Wei M, Lee C, Cohen P, Longo VD. Fasting and cancer treatment in humans: A case series report. Aging (Albany NY). 2009 Dec 31;1(12):988-1007. doi: 10.18632/aging.100114. PMID 20157582
- [Derived] Ligorio F, Lobefaro R, Fuca G, Provenzano L, Zanenga L, Nasca V, Sposetti C, Salvadori G, Ficchi A, Franza A, Martinetti A, Sottotetti E, Formisano B, Depretto C, Scaperrotta G, Belfiore A, Vingiani A, Ferraris C, Pruneri G, de Braud F, Vernieri C. Adding fasting-mimicking diet to first-line carboplatin-based chemotherapy is associated with better overall survival in advanced triple-negative breast cancer patients: A subanalysis of the NCT03340935 trial. Int J Cancer. 2024 Jan 1;154(1):114-123. doi: 10.1002/ijc.34701. Epub 2023 Aug 24. PMID 37615485
- [Derived] Ligorio F, Fuca G, Provenzano L, Lobefaro R, Zanenga L, Vingiani A, Belfiore A, Lorenzoni A, Alessi A, Pruneri G, de Braud F, Vernieri C. Exceptional tumour responses to fasting-mimicking diet combined with standard anticancer therapies: A sub-analysis of the NCT03340935 trial. Eur J Cancer. 2022 Sep;172:300-310. doi: 10.1016/j.ejca.2022.05.046. Epub 2022 Jul 8. PMID 35810555